CLINICAL TRIAL: NCT06125444
Title: IImpact of Hyperuricemia on Psoriatic Arthritis
Brief Title: Impact of Hyperuricemia on Psoriatic Arthritis
Acronym: Psoriatic
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 7957
Record Dates: First submitted 2022-11-14; First posted 2023-11-09 (Actual); Last update posted 2023-12-08 (Actual); Status verified 2023-12

CONDITIONS: Psoriatic Arthritis
Keywords: Psoriatic Arthritis; Hyperuricemia; Rheumatisms
MeSH Terms: conditions — Arthritis, Psoriatic; Hyperuricemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Psoriatic arthritis and gout (linked to hyperuricemia) are two rheumatisms well known to rheumatologists. There are epidemiological and physiopathological arguments in favor of a non-fortuitous link between these two rheumatisms, which to date has not been established. There is currently no recommendation to treat hyperuricaemia without an episode of gout attack. We hypothesize that there is a link between hyperuricemia and severity of rheumatism. This would ultimately modify the therapeutic management of hyperuricemic patients followed for psoriatic arthritis.

ELIGIBILITY:
Inclusion criteria:

* Major subject (≥18 years old)
* Subject with a history of psoriatic arthritis objectified according to the CIM 10-1 coding for patients followed in hospitalization at the HUS and HCC
* Subject presenting psoriatic arthritis objectified during a consultation by an HCC rheumatologist
* Among these two populations, all subjects for whom at least one serum uric acid assay was available in the medical file
* Subject having not expressed, after being informed, opposition to the reuse of their data for research purposes

Exclusion criteria:

* Subject who expressed their opposition to participating in the study
* Subject who met the inclusion criteria but whose analysis of the medical file (anamnestic, clinical, biological and radiological data) led to a diagnostic reversal and therefore did not present with psoriatic arthritis
* Subject under guardianship or curatorship
* Subject under safeguard of justice

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Major subject (≥18 years old), with a history of psoriatic arthritis objectified according to the CIM 10-1 coding for patients followed in hospitalization at the HUS and HCC and subject presenting psoriatic arthritis objectified during a consultation by an HCC rheumatologist
Sampling Method: Non-Probability Sample
Enrollment: 242 (Estimated)
Dates: Start 2020-08-24 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Retrospectively determine the impact of hyperuricemia on the response to psoriatic arthritis treatments: inventory of the latest treatments in progress and the response to treatment according to the treating rheumatologist | Files analysed retrospectively from January 01, 2009 to December 31, 2019 will be examined

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Rhumatologie - CHU de Strasbourg - France, Strasbourg, France